CLINICAL TRIAL: NCT00154128
Title: The Influence of of a Stabilization Splint on the Body Posture in TMD Cases and Controls
Brief Title: The Influence of a Stabilization Splint on the Body Posture
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RD-B-01
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-11-18 (Estimated); Status verified 2005-09

CONDITIONS: Temporomandibular Disorders; Craniomandibular Disorders; Arthromyalgia; Chronic Disease; Occlusal Appliance
Keywords: temporomandibular disorder; craniomandibular disorder; occlusal appliance; clinical trial
MeSH Terms: conditions — Temporomandibular Joint Disorders; Craniomandibular Disorders; Chronic Disease | interventions — Occlusal Splints

INTERVENTIONS:
Device: occlusal appliance

SUMMARY:
The study was designed to investigate a possible influence of an occlusal stabilization splint on the body posture in TMD cases and controls. Interocclusal appliances or occlusal splints are therapeutic devices that are most frequently used in the treatment of TMD. Changes of the mandibular position and occlusal equilibrations are assumed to have an impact on the general body posture.

DETAILED DESCRIPTION:
Thirty TMD cases and 10 controls were included in the study. All participants were recruited from the School of Dentistry, University of Greifswald. All subjects gave their written consent to participate in the study. They then completed a TMD history questionnaire and underwent a clinical examination. The examination included palpation of the masticatory muscles and the TMJs, range of mandibular motion measurements, and assessment of joint noises. The TMD cases were required to have a diagnoses of myofascial pain and/or arthralgia. Controls had to be free of pain symptoms in their masticatory muscles and TMJs. Body posture was measured during five minutes of walking using an ultrasound-distance measuring device (sonoSens® Monitor) with small sensors placed on the skin that continually record changes in the distance between them. A static posture evaluation was performed with a contactless, and radiation-free static measurement of the back surface and spine using a 3D measurement system (formetric II). A second measurement was performed after insertion of the occlusal appliance and a third one after 7 days of treatment.

The occlusal appliances were inserted after the first examination and all participants were instructed to use it at night and during examinations.

ELIGIBILITY:
Inclusion Criteria:

* TMD cases: diagnoses of myofascial pain and/or arthralgia

Exclusion Criteria:

* TMD cases: chronic systemic diseases, cardiac pacemakers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-04; Study Completion 2005-08

PRIMARY OUTCOMES:
changes in body posture

SECONDARY OUTCOMES:
score of compliants
number of tender muscles and TMJs

CONTACTS AND LOCATIONS:
Overall Officials: Georg Meyer, Prof., Principal Investigator — School of Dentistry, University of Greifswald, Germany; Georg Meyer, Prof. Dr., Principal Investigator — School of Dentistry, University of Greifswald